CLINICAL TRIAL: NCT00724230
Title: PegIntron/REBETOL Combination Therapy Designated Drug Use Investigation -Investigation on the Safety and Efficacy of PegIntron and REBETOL Combination Therapy in Patients With Chronic Hepatitis C Excluding Those With "IFN Naive Low Viral Load and Genotype 1 and High Viral Load"-
Brief Title: Safety and Efficacy of PegIntron Plus Rebetol in Patients With Chronic Hepatitis C in Japan, Excluding (1) Subjects With HCV Genotype 1 and High Viral Load, and (2) Interferon-naïve Subjects With Low Viral Load (Study P04841)(COMPLETED)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04841
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Hepatitis C, Chronic; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Arm 1: Overall study population.
  Interventions: Drug: PegIntron (peginterferon alfa-2b; SCH 54031); Drug: Rebetol (ribavirin; SCH 18908)

INTERVENTIONS:
Drug: PegIntron (peginterferon alfa-2b; SCH 54031) — PegIntron administered in accordance with approved labeling
  Subcutaneous injection once weekly for 24 weeks.
  Other Names: SCH 54031
Drug: Rebetol (ribavirin; SCH 18908) — Rebetol administered orally twice daily in accordance with approved labeling. Dosing duration 24 weeks.
  Other Names: SCH 18908

SUMMARY:
The objective of the study is to evaluate the safety and efficacy of PegIntron plus Rebetol combination therapy administered to patients with chronic hepatitis C. The study will exclude (1) subjects with HCV genotype 1 and high viral load, and (2) interferon-naïve subjects with low viral load. It is being conducted as a post-approval commitment, in accordance with the Ministry of Health, Labour and Welfare's guideline on Good Post-marketing Study Practice.

Post-marketing surveys are not considered applicable clinical trials and thus the results of this survey will not be posted at its conclusion. The results will be submitted to public health officials as required by applicable national and international laws.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with chronic hepatitis C
* Among interferon-naïve patients, only patients with high viral load and HCV genotype other than 1
* Among prior nonresponders or relapsers to interferon monotherapy, (1) patients with high viral load and HCV genotype other than 1; and (2) patients with low viral load of all genotypes (including genotype 1)

Exclusion Criteria:

* Patients infected with HCV genotype 1 with high viral load, regardless of whether treatment-naïve or previous nonresponders/relapsers
* Interferon-naïve patients with low viral load
* Patients with a history of hypersensitivity to test drugs or other interferon preparations
* Patients with a history of hypersensitivity to biological products, such as vaccines
* Patients being treated with Shosaikoto
* Patients with autoimmune hepatitis
* Pregnant women, women who may be pregnant, and nursing mothers
* Patients with a history of hypersensitivity to any component of this drug or other nucleoside analogs (aciclovir, ganciclovir, vidarabine, etc.)
* Patients with difficult-to-control cardiac disease (eg, myocardial infarction, cardiac failure, arrhythmia)
* Patients with hemoglobinopathies (eg, thalassemia, sickle-cell anemia)
* Patients with chronic renal failure or renal function disorder with creatinine clearance of <=50 mL/min
* Patients with or a history of severe psychiatric condition such as severe depression, suicidal ideation or suicide attempt
* Patients with serious hepatic dysfunction
* Patients with autoimmune hepatitis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with chronic hepatitis C excluding subjects with HCV genotype 1 and high viral load, and interferon-naïve subjects with low viral load. Patients undergoing treatment with PegIntron and Rebetol in clinical practice at approximately 50 to 100 sites in Japan.
Sampling Method: Non-Probability Sample
Enrollment: 505 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Overall incidence of adverse events and adverse drug reactions. | Assessed from the time the informed consent is signed up until 30 days after completion or discontinuation from the study
Assessment of trends of adverse drug reactions by patient factors and concomitant medications; Incidence, severity, and outcome of adverse events (AEs) between the elderly vs younger patients | Assessed from the time the informed consent is signed up until 30 days after completion or discontinuation from the study
Sustained virologic response rate by HCV genotype, baseline viral load, and patient demographic characteristics | Assessed at 24 weeks post-treatment

SECONDARY OUTCOMES:
Rate of ALT normalization at end of treatment period and at 24 weeks post completing therapy. | End of treatment and 24 weeks after end of treatment